CLINICAL TRIAL: NCT00197782
Title: The Immediate and Longterm Immune Responses of UK Infants and Young Children to a Booster Dose of Hib Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health England (Other Government)
Responsible Party: Principal Investigator, Prof. Elizabeth Miller, consultant epidemiologist, Public Health England
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Hibboost
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Haemophilus Influenzae Type b
MeSH Terms: conditions — Haemophilus Infections

INTERVENTIONS:
Biological: Hib conjugate vaccine

SUMMARY:
To measure the magnitude and persistence of the antibody response to a booster dose of Hib conjugate vaccine given between 9 months and 4 years of age to UK children who had completed primary immunisation with 3 doses of Hib vaccine given at 2/3/4 months of age either as a combined D/T/wholecellpertussis/Hib or D/T/acellularpertussis/Hib vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from parent or legal guardian of the infant or child
* Age >= 9 months and <4 years at recruitment
* Eligible to receive a single dose of Hib vaccine as per the UK schedule
* Receipt of three doses of Hib vaccine in infancy

Exclusion Criteria:

* History of Hib infection
* History of severe local reaction that can be confidently related to a prior Hib immunisation
* Deferral of vaccination if acute illness and/or temperature >38C on day of vaccination

Ages: 9 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2003-04; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MBBS FRCPath, Principal Investigator — Public Health England

REFERENCES:
- [Result] Southern J, McVernon J, Gelb D, Andrews N, Morris R, Crowley-Luke A, Goldblatt D, Miller E. Immunogenicity of a fourth dose of Haemophilus influenzae type b (Hib) conjugate vaccine and antibody persistence in young children from the United Kingdom who were primed with acellular or whole-cell pertussis component-containing Hib combinations in infancy. Clin Vaccine Immunol. 2007 Oct;14(10):1328-33. doi: 10.1128/CVI.00191-07. Epub 2007 Aug 15. PMID 17699835